CLINICAL TRIAL: NCT04032652
Title: Measurement of Rectal Levels of 5-aminosalicylic Acid (5-ASA) Using a Novel In-vivo Rectal Dialysis Technique in Healthy Volunteers on Asacol
Brief Title: Use of Rectal Dialysis Technique to Measure Rectal 5-ASA Levels in Healthy Volunteers Receiving Asacol
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Insufficient enrollment
Sponsor: Endeavor Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: EH 11-364
Record Dates: First submitted 2012-12-04; First posted 2019-07-25 (Actual); Results first posted 2019-10-15 (Actual); Last update posted 2019-10-15 (Actual); Status verified 2019-09

CONDITIONS: Ulcerative Colitis
Keywords: Pharmacokinetics; Aminosalicylates; Mucosal levels; Rectal dialysis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1200 mg Asacol once daily for 1 week (Active Comparator): Rectal dialysis will be done after 1 week on 1200 mg asacol
  Interventions: Procedure: Rectal dialysis; Drug: Rectal dialysis
- 2400 mg Asacol once daily for 1 week (Active Comparator): Rectal dialysis will be done after 1 week on 2400 mg asacol
  Interventions: Procedure: Rectal dialysis; Drug: Rectal dialysis

INTERVENTIONS:
Procedure: Rectal dialysis — Rectal dialysis done after 1 week on either 1200/2400 mg Asacol dose to test rectal mucosal 5-ASA levels
Drug: Rectal dialysis — Rectal dialysis done after 1 week on either 1200/2400 mg Asacol dose to test rectal mucosal 5-ASA levels

SUMMARY:
The investigators plan to develop a novel method of estimating 5-ASA levels in the rectum at a mucosal level using in vivo rectal dialysis technique towards the eventual goal of determining the optimal dosing of Asacol® that would provide therapeutic levels of 5-ASA in the left colon.

DETAILED DESCRIPTION:
Asacol® is mesalazine in a pH-dependent tablet (Eudragit S) that remains intact until reaching the terminal ileum. The tablet dissolves at a pH 7 or greater, allowing mesalazine release in the terminal ileum and throughout the colon; hence, it would be anticipated that this form of 5-ASA will produce higher concentrations in the left colon in patients with active ulcerative colitis compared to other immediate release forms of 5-ASA. However, preliminary research using dynamic computer modeling and simulation predicted that patients with active ulcerative colitis (characterized by an increased stool frequency) treated with Asacol® and Lialda (another delayed release formulation) will achieve very low 5-ASA levels in the sigmoid colon and rectum. The model predicts that these 5-ASA preparations will be relatively ineffective in treating the left side of the colon in active ulcerative colitis.

ELIGIBILITY:
Inclusion Criteria:

* Eligible subjects would be healthy males and females
* 18-45 years of age (inclusive)
* Within 20% of normal body weight at screening
* Who are able to give written informed consent.

Exclusion Criteria:

* History of any chronic illness
* Evidence of significant organic or psychiatric disease on a brief health questionnaire
* A history or presence of any condition causing malabsorption or an effect on gastrointestinal motility
* A history of any gastrointestinal surgery
* A history of acute or chronic renal insufficiency
* Pre existing liver disease
* A history of severe allergic reaction to salicylates, aminosalicylates or any of the ingredients of Asacol® tablets or a history of multiple food/drug allergies or if they are pregnant or lactating.
* Subjects will be required to refrain from any prescription or nonprescription drug or herbal products except their birth control medications for gastrointestinal disorders for 7 days prior to dosing and during the study, till its completion at the end of the fifth visit.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2 (Actual)
Dates: Start 2012-12 (Actual); Primary Completion 2014-11 (Actual); Study Completion 2014-12-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eli D Ehrenpreis, MD, Principal Investigator — Endeavor Health

REFERENCES:
- [Background] Stobaugh DJ, Deepak P, Thorpe M, Hannon B, Ehrenpreis ED. Simulated comparison of topical and oral formulations of 5-aminosalicylate for the treatment of ulcerative colitis. Inflamm Bowel Dis. 2013 Feb;19(2):301-8. doi: 10.1002/ibd.23003. PMID 22644716
- [Background] Reissman P, Ehrenpreis ED, Cohen S, Nogueras JJ, Zaitman D, Wexner SD. Electrolyte profiles within the ileoanal pouch: measurement by an in vivo equilibrium dialysis technique. Dig Liver Dis. 2003 Apr;35(4):251-5. doi: 10.1016/s1590-8658(03)00062-8. PMID 12801036

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study was terminated and the PI has left the institution. Efforts were made to contact the PI/study team members, but were unsuccessful. No study data are available.
Period: Overall Study
Arm/Group | 1200 mg Asacol Once Daily for 1 Week | 2400 mg Asacol Once Daily for 1 Week
Started | 1 | 1
Completed | 0 | 0
Not Completed | 1 | 1
Not completed — The study was terminated and the PI has | 1 | 1

BASELINE CHARACTERISTICS:
Population: The study was terminated and the PI has left the institution. Efforts were made to contact the PI/study team members, but were unsuccessful. No study data are available
Groups:
- Total: Total of all reporting groups
Arm/Group | 1200 mg Asacol Once Daily for 1 Week | 2400 mg Asacol Once Daily for 1 Week | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Categorical
Age, Continuous
Sex: Female, Male
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Detection of 5-ASA
Description: 5-ASA to be measured using rectal dialysis technique in-vivo
Time Frame: 2 weeks after starting Asacol
Population: as for baseline characteristics
Arm/Group | 1200 mg Asacol Once Daily for 1 Week | 2400 mg Asacol Once Daily for 1 Week
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Change in Detected 5-ASA With Change in Ingested Asacol Dose
Description: Comparison of 2-week and 5-week 5-ASA as measured thorugh rectal dialysis
Time Frame: 5 weeks after starting study
Population: as for baseline characteristics
Arm/Group | 1200 mg Asacol Once Daily for 1 Week | 2400 mg Asacol Once Daily for 1 Week
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: The study was terminated and the PI has left the institution. Efforts were made to contact the PI/study team members, but were unsuccessful. No study data are available, including data about adverse events.
Arm/Group | 1200 mg Asacol Once Daily for 1 Week | 2400 mg Asacol Once Daily for 1 Week
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
The study was terminated and the PI has left the institution. Efforts were made to contact the PI/study team members, but were unsuccessful. No study data are available

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes